CLINICAL TRIAL: NCT02365727
Title: Two-arm, Double-blind Randomized Study Comparing Exparel and Exparel Plus an Adductor Canal Block in Total Knee Arthroplasty
Brief Title: Exparel vs Exparel Plus ACB in TKAs
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol not feasible as written
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00034356
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine; Epinephrine; Clonidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exparel plus Adductor Canal Block (Experimental): Adductor canal block with 20 cc 0.5% Ropivacaine with 1:400,000 epinephrine and 100mcg of clonidine
  Interventions: Drug: Liposomal bupivacaine; Drug: Ropivacaine; Drug: Epinephrine; Drug: Clonidine
- Exparel plus Placebo Block (Placebo Comparator): Adductor canal block with 20 cc saline
  Interventions: Drug: Liposomal bupivacaine; Drug: Saline

INTERVENTIONS:
Drug: Liposomal bupivacaine
  Other Names: Exparel
Drug: Ropivacaine
  Arms: Exparel plus Adductor Canal Block
Drug: Epinephrine
  Arms: Exparel plus Adductor Canal Block
Drug: Clonidine
  Arms: Exparel plus Adductor Canal Block
Drug: Saline
  Arms: Exparel plus Placebo Block

SUMMARY:
Patients will be randomized (like the flip of a coin) to receive Exparel and a nerve block, standard of care for this procedure, or Exparel alone for pain management after surgery. They will also be asked to complete questionnaires before surgery, during their stay at the hospital after surgery, then at 3 months, 6 months and 12 months after surgery to assess pain and/or function levels, as well as the amount of pain medicine patients have used after surgery. Patients' leg strength will be measured immediately after surgery and again at 3, 6 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 80 years at the time of surgery.
* Willing and able to give voluntary informed consent to participate in this investigation.
* Candidate for total knee arthroplasty.
* BMI < 35.

Exclusion Criteria:

* Subject has had previous arthroplasty or fracture procedure(s) on the operative knee.
* Creatine level ≥ 1.5
* Pre-existing gait disturbance or neuropathy.
* Allergy to local anesthetics.
* Inflammatory arthropathies.
* Female patient who is pregnant or nursing.
* Chronic use of narcotics
* Any other reason (in the judgment of the investigator).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain as assessed by Visual Analog Scale (VAS) | 12 Months
  Pain, as assessed by Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Function as assessed by Knee Society Score (KSS) and EQ-5D | 12 Months
  Function, as assessed by Knee Society Score (KSS) and EQ-5D
Opioid consumption as assessed by dosage and frequency of narcotic usage | 30 hours
  Opioid consumption, as assessed by dosage and frequency of narcotic usage

CONTACTS AND LOCATIONS:
Overall Officials: Brayton Shirley, Principal Investigator — Steadman Hawkins Clinic of the Carolinas - Greenville Health System
Locations (1):
- Steadman Hawkins Clinic of the Carolinas - Greenville Health System, Greenville, South Carolina, United States